CLINICAL TRIAL: NCT03718884
Title: Evaluation of the Effect of Mirikizumab on the Pharmacokinetics of Cytochrome P450 Substrates in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Mirikizumab in Participants With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17117; I6T-MC-AMBP (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Cocktail (Experimental): Period 1:
  Participants received a single dose of the following drug cocktail on Day 1: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg Caffeine administered orally
  Interventions: Drug: Drug Cocktail
- Mirikizumab + Drug Cocktail (Experimental): Period 2:
  Participants received 250 mg mirikizumab subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks (Days 1 to Day 113)
  Period 2:
  Participants received the second dose of the drug cocktail: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg caffeine administered orally on Day 116.
  Interventions: Drug: Drug Cocktail; Drug: Mirikizumab

INTERVENTIONS:
Drug: Drug Cocktail — Drug cocktail consists of caffeine, warfarin plus vitamin K, omeprazole, dextromethorphan, and midazolam, administered orally
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab + Drug Cocktail

SUMMARY:
This study is known as a "drug interaction study." The purpose is to learn how commonly used drugs or substances (midazolam, warfarin, dextromethorphan, omeprazole, and caffeine) and their breakdown products get into the bloodstream after taking a "cocktail" (combination) of them before and after multiple doses of mirikizumab.

The study will last about 23 weeks for each participant. Screening must be completed within 4 weeks prior to study start.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with chronic plaque psoriasis for at least 6 months who are candidates for systemic therapy or phototherapy
* Have greater than or equal to (≥) 10 percent body surface area (BSA) involvement at screening and first admission to the clinical site

Exclusion Criteria:

* Pregnant or nursing (lactating)
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection
* Have major surgery within 8 weeks prior to first admission to the clinical site or during the study
* Have a history of lymphoma, leukemia, or any malignancy
* Require treatment with the cocktail drugs within 14 days prior to the first administration of the drug cocktail through the end of Week 12 assessments
* Have participated in any other study with mirikizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Avail Clinical Research LLC, DeLand, Florida
  - High Point Clinical Trials Center, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirikizumab + Drug Cocktail: Period 2:
  Participants received 250 mg mirikizumab subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks (Days 1 to Day 113).
  Period 2:
  Participants received the second dose of the drug cocktail: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg caffeine administered orally on Day 116.
Period: Period 1 (6 Days)
Arm/Group | Drug Cocktail | Mirikizumab + Drug Cocktail
Started | 29 | 0 (Participants were assigned to this arm only during Period 2.)
Received at Least One Dose of Study Drug | 29 | 0
Completed | 29 | 0 (Participants were assigned to this arm only during Period 2.)
Not Completed | 0 | 0
Period: Period 2 (120 Days)
Arm/Group | Drug Cocktail | Mirikizumab + Drug Cocktail
Started | 0 (Participants were assigned to this arm only during Period 1.) | 29 (Participants were assigned to this arm only during Period 2.)
Completed | 0 (Participants were assigned to this arm only during Period 1.) | 26
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Drug Cocktail
  Period 1:
  Participants received a single dose of the following drug cocktail on Day 1: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg Caffeine administered orally.
  Mirikizumab + Drug Cocktail
  Period 2:
  Participants received 250 mg mirikizumab subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks (Days 1 to Day 113)
  Period 2:
  Participants received the second dose of the drug cocktail: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg caffeine administered orally on Day 116.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 52.1 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Midazolam
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Midazolam
Time Frame: Period 1: Day 1: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 2: 24 hours; Period 2: Day 116: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 117: 24 hours; post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilitre (ng/mL)
Groups:
- Period 1: 1 mg Midazolam: Period 1: Participants received 1 mg midazolam administered orally on Day 1.
- Period 2: 1 mg Midazolam: Period 2: Participants received 1 mg midazolam administered orally on day 116.
Arm/Group | Period 1: 1 mg Midazolam | Period 2: 1 mg Midazolam
Number analyzed (Participants) | 29 | 26
Nanograms per millilitre (ng/mL) | 4.07 (29) | 4.46 (35)

2. Primary Outcome: PK: Cmax of Warfarin
Description: PK: Cmax of Warfarin
Time Frame: Period 1: Day 1: predose,1,2, 4,6, 8 and 10 hours, Day 2: 24 hours, Day 3: 48 hours, Day 4: 72 hours, Day 5: 96 hours; Period 2: Day 116: predose,1,2,4,6,8 and 10 hours, Day 117: 24 hours, Day 118: 48 hours, Day 119: 72 hours, Day 120: 96 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1: 10 mg Warfarin: Period 1: Participants received 10 mg warfarin administered orally on Day 1.
- Period 2: 10 mg Warfarin: Period 2: Participants received 10 mg warfarin administered orally on day 116.
Arm/Group | Period 1: 10 mg Warfarin | Period 2: 10 mg Warfarin
Number analyzed (Participants) | 29 | 26
ng/mL | 543 (18) | 506 (23)

3. Primary Outcome: PK: Cmax of Dextromethorphan
Description: PK: Cmax of Dextromethorphan
Time Frame: Period 1: Day 1: predose, 1, 2, 4, 6, 8 and 10 hours, Day 2: 24 hours, Day 3: 48 hours, Day 4: 72 hours; Period 2: Day 116: predose, 1, 2,4, 6, 8 and 10 hours, Day 117: 24 hours, Day 118: 48 hours, Day 119: 72 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1: 30 mg Dextromethorphan: Period 1: Participants received 30 mg dextromethorphan administered orally on Day 1.
- Period 2: 30 mg Dextromethorphan: Period 2: Participants received 30 mg dextromethorphan administered orally on day 116.
Arm/Group | Period 1: 30 mg Dextromethorphan | Period 2: 30 mg Dextromethorphan
Number analyzed (Participants) | 29 | 26
ng/mL | 1.60 (154) | 1.47 (118)

4. Primary Outcome: PK: Cmax of Omeprazole
Description: PK: Cmax of Omeprazole
Time Frame: Period 1: Day 1: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 2: 24 hours, Day 3: 48 hours; Period 2: Day 116: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 117: 24 hours, Day 118: 48 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1: 20 mg Omeprazole: Period 1: Participants received 20 mg omeprazole administered orally on Day 1.
- Period 2: 20 mg Omeprazole: Period 2: Participants received 20 mg omeprazole administered orally on day 116.
Arm/Group | Period 1: 20 mg Omeprazole | Period 2: 20 mg Omeprazole
Number analyzed (Participants) | 29 | 26
ng/mL | 369 (137) | 437 (81)

5. Primary Outcome: PK: Cmax of Caffeine
Description: PK: Cmax of Caffeine
Time Frame: as for outcome 4
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1: 100 mg Caffeine: Period 1: Participants received 100 mg caffeine administered orally on Day 1.
- Period 2: 100 mg Caffeine: Period 2: Participants received 100 mg caffeine administered orally on day 116.
Arm/Group | Period 1: 100 mg Caffeine | Period 2: 100 mg Caffeine
Number analyzed (Participants) | 26 | 18
ng/mL | 2400 (19) | 2340 (26)

6. Primary Outcome: PK: Area Under the Concentration Curve (AUC) Time Zero to Infinity (AUC [0-∞]) of Midazolam
Description: PK: Area Under the Concentration Curve (AUC) Time Zero to Infinity (AUC [0-∞]) of Midazolam
Time Frame: Period 1: Day 1: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 2: 24 hours; Period 2: Day 116: predose, 0.5, 1, 2, 3, 4, 6, 8 and 12 hours, Day 117: 24 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms hour per millilitre (ng*h/mL)
Arm/Group | Period 1: 1 mg Midazolam | Period 2: 1 mg Midazolam
Number analyzed (Participants) | 29 | 26
Nanograms hour per millilitre (ng*h/mL) | 13.4 (43) | 15.6 (40)

7. Primary Outcome: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Warfarin
Description: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Warfarin
Time Frame: Period 1: Day 1: predose,1,2,4,6,8 and 10 hours, Day 2: 24 hours, Day 3: 48 hours, Day 4: 72 hours, Day 5: 96 hours; Period 2: Day 116: predose, 1, 2, 4, 6, 8 and 10 hours, Day 117: 24 hours, Day 118: 48 hours,Day 119: 72 hours,Day 120: 96 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 1: 10 mg Warfarin | Period 2: 10 mg Warfarin
Number analyzed (Participants) | 28 | 25
ng*h/mL | 14800 (34) | 13800 (31)

8. Primary Outcome: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Dextromethorphan
Description: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Dextromethorphan
Time Frame: Period 1: Day 1: predose,1,2,4,6,8 and 10 hours, Day 2: 24 hours, Day 3: 48 hours, Day 4: 72 hours; Period 2: Day 116: predose, 1, 2,4, 6, 8 and 10 hours, Day 117: 24 hours, Day 118: 48 hours, Day 119: 72 hours;post-dose
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 1: 30 mg Dextromethorphan | Period 2: 30 mg Dextromethorphan
Number analyzed (Participants) | 29 | 26
ng*h/mL | 14.6 (160) | 13.0 (132)

9. Primary Outcome: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Omeprazole
Description: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Omeprazole
Time Frame: as for outcome 4
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 1: 20 mg Omeprazole | Period 2: 20 mg Omeprazole
Number analyzed (Participants) | 20 | 20
ng*h/mL | 1280 (142) | 1530 (103)

10. Primary Outcome: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Caffeine
Description: PK: AUC Time Zero to Infinity (AUC[0-∞]) of Caffeine
Time Frame: as for outcome 4
Population: All participants who received at least one dose of study drug cocktail and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 1: 100 mg Caffeine | Period 2: 100 mg Caffeine
Number analyzed (Participants) | 24 | 18
ng*h/mL | 19700 (46) | 20800 (48)

ADVERSE EVENTS:
Time Frame: Baseline Up To 144 Days
Description: All Participants who received at least one dose of study drug.
Groups:
- Period 1: Drug Cocktail: Period 1:
  Participants received a single dose of the following drug cocktail on Day 1: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg Caffeine administered orally.
- Period 2: Mirikizumab: Period 2:
  Participants received 250 mg mirikizumab subcutaneously (SC) once every 4 weeks (Q4W) for 16 weeks (Days 1 to Day 113).
- Period 2: Drug Cocktail: Period 2:
  Participants received the second dose of the drug cocktail: 1 mg midazolam, 10 mg warfarin, 10 mg vitamin K, 30 mg dextromethorphan, 20 mg omeprazole, 100 mg caffeine administered orally on Day 116.
Arm/Group | Period 1: Drug Cocktail | Period 2: Mirikizumab | Period 2: Drug Cocktail
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 3/29 | 0/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Drug Cocktail (N=29) | Period 2: Mirikizumab (N=29) | Period 2: Drug Cocktail (N=29)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT03718884/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT03718884/SAP_001.pdf